CLINICAL TRIAL: NCT06327594
Title: Study on the Value of Musculoskeletal Cross-modal Imaging Assessment System in the Diagnosis and Prognosis of Sarcopenia in Lung Cancer Patients
Brief Title: Assessment System of Sarcopenia in Lung Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xinyi Tang, Principal Investigator, West China Hospital
Other Study IDs: XTang-0002
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Sarcopenia; Lung Cancer; Ultrasound
MeSH Terms: conditions — Sarcopenia; Lung Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung cancer patients with sarcopenia
  Interventions: Diagnostic Test: ultrasound scan; Diagnostic Test: CT/MRI scan
- Lung cancer patients without sarcopenia
  Interventions: Diagnostic Test: ultrasound scan; Diagnostic Test: CT/MRI scan

INTERVENTIONS:
Diagnostic Test: ultrasound scan — The patients with lung cancer who are scheduled to undergo radical resection of lung cancer are examined by ultrasound at multiple sites of the whole body, including muscle and fat.
Diagnostic Test: CT/MRI scan — The patients with lung cancer who are scheduled to undergo radical resection of lung cancer are examined by abdominal CT/MRI.

SUMMARY:
1. To explore the diagnostic value of musculoskeletal cross-modal imaging assessment system of ultrasound combined with abdominal CT/MRI for sarcopenia in patients with lung cancer.
2. To explore the value of musculoskeletal cross-modal imaging assessment system of ultrasound combined with abdominal CT/MRI in evaluating the prognosis and the effect of nutritional support in patients with lung cancer during perioperative period.
3. To explore the value of musculoskeletal cross-modal imaging assessment system of ultrasound combined with abdominal CT/MRI in evaluating the long-term prognosis of patients with lung cancer.

DETAILED DESCRIPTION:
Sarcopenia is a progressive and systemic skeletal muscle disease that involves accelerated loss of muscle mass and function and is associated with increased adverse outcomes in older adults such as falls, functional decline, weakness, and death. It can be comorbid with a variety of diseases and interacts extensively with various disease states to influence disease prognosis. According to literature reports, the prevalence of sarcopenia in lung cancer patients is 42.8%-45.0%, and many studies have confirmed that sarcopenia is associated with a variety of poor prognosis of lung cancer. Early identification of sarcopenia in lung cancer patients and early intervention before the surgery are very important steps to improve the prognosis of lung patients.

However, at present, the evaluation methods of sarcopenia are very complicated, which rely on three features: loss of muscle mass, loss of muscle strength, and loss of physical performance. At present, physicians usually use bioelectrical impedance analysis (BIA) or dual-energy X-ray absorptiometry (DXA) to determine skeletal muscle mass index SMI to measure muscle mass, grip strength test to measure muscle strength, gait speed or tools such as SPPB scores to assess physical performance. A diagnosis of sarcopenia can be made when a subject experiences a decrease in SMI combined with a decrease in grip strength or a decrease in gait speed. The above evaluation methods are difficult to be used as routine preoperative evaluation items.

Previous studies have demonstrated that SMI in older adults can be accurately estimated by using muscle thickness acquired from ultrasound examination with basic information such as age and body mass index (BMI). And it has been shown that the cross-sectional area of the psoas major muscle at L3-level assessed by CT/MRI can also preliminarily diagnose sarcopenia. However, existing alternatives for assessing sarcopenia with ultrasound or CT/MRI alone are incomplete and lack stability.

Fronted with such a dilemma, we attempted to establish a musculoskeletal cross-modal imaging evaluation system of ultrasound combined with abdominal CT/MRI images, which can diagnose sarcopenia more comprehensively and accurately, and evaluate the perioperative prognosis, nutritional support effect and long-term prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients scheduled for radical resection of lung cancer.
2. With a CT/MRI examination within 1 week.
3. The compliance of examination was good.

Exclusion Criteria:

1. Amputated arm or leg.
2. Severe oedema (oedema higher than knee level).
3. Implantable pacemaker.
4. Impaired consciousness, poor general health, or other reasons that would prevent the individual from completing the study.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients scheduled for radical resection of lung cancer.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Death | Within 2 years after the initial ultrasound examination
Perioperative complications | Within 7 days after the surgery.
  Including local incision complications (infection, dehiscence); atelectasis/pulmonary infection; urinary tract infections; postoperative bleeding; deep venous thrombosis of the lower extremity; urinary retention; sepsis; hypoproteinemia, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xinyi Tang, Principal Investigator — Department of Medical Ultrasound, West China Hospital, Sichuan University
Locations (1):
- Xinyi Tang, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
By submitting an application to the project leader via email and obtaining approval from relevant hospital departments.